CLINICAL TRIAL: NCT00001338
Title: A Prospective, Randomized, Phase III Trial of FLAC (5-Fluorouracil, Leucovorin, Adriamycin, Cytoxan) Chemotherapy With GM-CSF (Granulocyte-Macrophage Colony-Stimulating Factor) Versus PIXY 321 in Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 930153; 93-C-0153
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-04

CONDITIONS: Breast Neoplasms; Fever; Hematologic Diseases; Neutropenia; Sepsis
Keywords: Fusion Protein
MeSH Terms: conditions — Breast Neoplasms; Fever; Hematologic Diseases; Neutropenia; Sepsis | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

INTERVENTIONS:
Drug: FLAC chemotherapy with GM-CSF

SUMMARY:
This is a prospective, randomized Phase III trial of FLAC chemotherapy with GM-CSF versus PIXY321 in advanced breast cancer. The primary endpoints of this study will be the duration of thrombocytopenia and the time to recovery of platelets to 50,000/microliters. Other clinical endpoints will include the depth and duration of leukopenia, neutropenia, and anemia, the platelet and RBC transfusion requirements, and the number of documented instances of sepsis and hospitalizations for fever and neutropenia.

Laboratory correlates will include the detailed evaluation of the effects on circulating hematopoietic progenitor cells by GM-CSF and PIXY321 and the potential effects these agents have on the bone marrow micro-environment.

After 5 cycles of FLAC with GM-CSF versus PIXY321, patients will be treated with 5 cycles of 96 hour infusional taxol. The goal of this part of the study will be to assess the toxicity and feasibility of administering infusional taxol following dose-intensive FLAC chemotherapy.

DETAILED DESCRIPTION:
This is a prospective, randomized Phase III trial of FLAC chemotherapy with GM-CSF versus PIXY321 in advanced breast cancer. The primary endpoints of this study will be the duration of thrombocytopenia and the time to recovery of platelets to 50,000/microliters. Other clinical endpoints will include the depth and duration of leukopenia, neutropenia, and anemia, the platelet and RBC transfusion requirements, and the number of documented instances of sepsis and hospitalizations for fever and neutropenia.

Laboratory correlates will include the detailed evaluation of the effects on circulating hematopoietic progenitor cells by GM-CSF and PIXY321 and the potential effects these agents have on the bone marrow micro-environment.

After 5 cycles of FLAC with GM-CSF versus PIXY321, patients will be treated with 5 cycles of 96 hour infusional taxol. The goal of this part of the study will be to assess the toxicity and feasibility of administering infusional taxol following dose-intensive FLAC chemotherapy.

ELIGIBILITY:
Patients with Stage IV (metastatic) breast cancer who have a histologically-proven diagnosis. Measurable, evaluable Stage III patients, Stage II patients with 4 or more nodes positive, and Stage IV NED (no evidence of disease) patients.

Patients who have had prior radiation therapy providing there was not more than 20% of the bone marrow has been irradiated.

Patients who have received less than or equal to 360mg/m2 of Adriamycin as adjuvant therapy.

Patients must be previously untreated with chemotherapy for metastatic disease.

There must be no history of previous malignancy except for cured non-melanoma skin cancer (basal or squamous cell carcinoma), cervical cancer in situ, or a past malignancy that has been inactive for over 5 years.

Performance status (Karnofsky scale) must be greater than 70; ECOG 0-2.

Absolute granulocyte count greater than 1500 microliters and platelet count greater than 100,000/mm3.

Liver function tests (SGOT, and total bilirubin) should be less than 2X the upper limits of normal unless there is evidence of hepatic involvement with tumor. Serum creatinine should be less than 1.7 or creatinine clearance should be greater than 45 ml/min.

Patients must be greater than or equal to 18 years of age.

The patient must be able to give informed consent, and to return to NCI for treatment and adequate follow-up for the period the protocol requires.

No patients who are poor medical or psychiatric risks because of nonmalignant systemic disease which would preclude them from being subjected to any treatments in this protocol.

Patients should not currently require therapy for cardiac arrhythmias, congestive heart failure, or coronary artery disease. Patients who have received prior Adriamycin or have any history of cardiac disease must have a LVEF greater than 45 percent by MUGA.

No history of CNS metastasis, or know seizure disorder.

No allergy to any study medication.

No pregnant or lactating women.

No patients requiring ongoing therapy for asthma.

No patients with bleeding disorders for study entry as are patients requiring chronic anticoagulation.

No patients with active infection or are known to be HIV positive.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65
Dates: Start 1993-06; Study Completion 2001-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Horton JK, Thimmaiah KN, Houghton JA, Horowitz ME, Houghton PJ. Modulation by verapamil of vincristine pharmacokinetics and toxicity in mice bearing human tumor xenografts. Biochem Pharmacol. 1989 Jun 1;38(11):1727-36. doi: 10.1016/0006-2952(89)90405-x. PMID 2735930
- [Background] Lai GM, Chen YN, Mickley LA, Fojo AT, Bates SE. P-glycoprotein expression and schedule dependence of adriamycin cytotoxicity in human colon carcinoma cell lines. Int J Cancer. 1991 Nov 11;49(5):696-703. doi: 10.1002/ijc.2910490512. PMID 1682280
- [Background] Buzzoni R, Bonadonna G, Valagussa P, Zambetti M. Adjuvant chemotherapy with doxorubicin plus cyclophosphamide, methotrexate, and fluorouracil in the treatment of resectable breast cancer with more than three positive axillary nodes. J Clin Oncol. 1991 Dec;9(12):2134-40. doi: 10.1200/JCO.1991.9.12.2134. PMID 1960555